CLINICAL TRIAL: NCT00320151
Title: Collection of Blood for Gene Expression Study in Individuals With Chronic Lung Diseases
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: Blood Collection Protocol
Record Dates: First submitted 2006-04-27; First posted 2006-05-03 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Diseases
Keywords: chronic lung disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol is designed to gather a small amount of blood from patients seen in the New York Presbyterian Hospital-Weill Cornell Medical Center Pulmonary, Critical Care unit, and 5 West floor (Pulmonary Floor) for clinical care associated with chronic lung disease. This protocol will also survey medical records of patients with chronic lung disease, in order to study the clinical characteristics of these individuals. Investigators aim to understand the genetics of chronic lung diseases, and will use the serum and DNA from this blood to perform various genotyping studies such as such as genomic/gene expression studies of individuals with chronic lung diseases

DETAILED DESCRIPTION:
This protocol is designed to gather a small amount of blood from patients seen in the New York Presbyterian Hospital-Weill Cornell Medical Center Pulmonary, Critical Care unit, and 5 West floor (Pulmonary Floor) for clinical care associated with chronic lung disease. This protocol will also survey medical records of patients with chronic lung disease, in order to study the clinical characteristics of these individuals. Investigators aim to understand the genetics of chronic lung diseases, and will use the serum and DNA from this blood to perform various genotyping studies such as such as genomic/gene expression studies of individuals with chronic lung diseases.

General admission criteria for this project will require at least one of the following: (1) symptoms consistent with pulmonary disease; (2) chest X-ray consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and (6) patients with diseases of organs with known association with lung disease.

The following studies will be conducted on blood specimens: genomic DNA will be extracted; promoter sequences for antioxidant-related genes will be obtained by PCR and sequenced. The goal is to find single nucleotide polymorphisms (SNP) to see if they correlate with lung disease. DNA samples and blood specimens will be coded. Samples could potentially be traced back to the patient. However, every effort will be made to keep the patient's identity confidential per HIPAA regulations.

The study does not aim to create a blood bank. Rather, the blood samples will be used for DNA extraction only. Serum will be stored for future studies, to look at levels of proteins.

ELIGIBILITY:
Inclusion Criteria:

* Must provide informed consent
* Males and females, age 18 years and older
* Lung disease proven by at least one of the following: (1) symptoms consistent with pulmonary disease; (2) chest X-rays consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and (6) diseases of organs with known association with lung disease

Exclusion Criteria:

* Drug and/or alcohol abuse within the past six months
* Females who are pregnant or nursing

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General admission criteria for this project will require at least one of the following: (1) symptoms consistent with pulmonary disease; (2) chest X-ray consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and (6) patients with diseases of organs with known association with lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 3087 (Actual)
Dates: Start 2006-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Crystal, M.D., Principal Investigator — Weill Medical College of Cornell University; Ben-Gary Harvey, M.D., Study Director — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided